CLINICAL TRIAL: NCT03854435
Title: Determination of Heart Rate in Infants Needing Resuscitation at Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Padova (Other)
Collaborators: CUAMM Doctors with Africa, Padova, Italy (Unknown); St. Luke Catholic Hospital, Wolisso, Ethiopia (Unknown)
Responsible Party: Principal Investigator, Daniele Trevisanuto, Professor, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: University of Padova
Record Dates: First submitted 2019-01-29; First posted 2019-02-26 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Perinatal Asphyxia
MeSH Terms: interventions — Stethoscopes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart rate assessed by using a stethoscope (auscultation) (Experimental): Heart rate will be assessed by using a stethoscope (auscultation) in newborn infants immediately after birth
  Interventions: Other: Heart rate assessment (stethoscope)
- Heart rate assessed by palpation of the umbilical cord (Active Comparator): Heart rate will be assessed by palpation of the umbilical in newborn infants immediately after birth
  Interventions: Other: Heart assessment (umbilical cord palpation)

INTERVENTIONS:
Other: Heart rate assessment (stethoscope) — Immediately after birth heart rate will be evaluated by auscultation
  Arms: Heart rate assessed by using a stethoscope (auscultation)
Other: Heart assessment (umbilical cord palpation) — Immediately after birth heart rate will be evaluated by palpation of the umbilical cord
  Arms: Heart rate assessed by palpation of the umbilical cord

SUMMARY:
Algorithms for neonatal resuscitation adapted to low resource settings include HR evaluation by auscultation or umbilical cord palpation at about one minute of life.

Previous studies conducted in high resource settings showed that auscultation of the precordium is more accurate than umbilical palpation to assess HR of healthy infants at birth.The last versions of the American Heart Association and the European Resuscitation Council Guidelines on Neonatal resuscitation suggest that "during resuscitation of term and preterm newborns, the use of 3-lead ECG for the rapid and accurate measurement of the newborn's heart rate may be reasonable". However, this remains a weak recommendation with a very-low-quality evidence.

In low resource countries, a stethoscope is rarely available and palpation of the umbilical pulse is the method used for detecting HR. Although this is preferable to other palpation sites (i.e. femo-ral and brachial artery), there is a high likelihood of underestimating HR with palpation of the umbilical pulse in healthy infants.

The accuracy of assessing HR by auscultation and umbilical palpation in newborn infants requir-ing resuscitation remains unknown.

To the investigator's knowledge, there are not previous studies that have compared the accuracy of HR estima-tion by auscultation vs. umbilical palpation in newborn infants needing resuscitation This study was designed to compare two different methods (auscultation and umbilical cord pal-pation) of HR estimation in newborn infants needing resuscitation, in order to determine which method is most suitable for use in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. inborn infants (and)
2. need for resuscitation (and)
3. parental consent; a written informed consent will be obtained by a member of the neonatal staff involved in the study from a parent or guardian at maternal admission to the obstetrical ward or prior to delivery.

Exclusion Criteria:

1. Major congenital malformations;
2. Parental refusal to participate to the study.

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Meles and females will be enrolled
Enrollment: 60 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Degree of agreement of herat rate obtained by auscultation or palpation (HR: <60bpm/60-100bpm/>100bpm) obtained by auscultation or palpation compared with the HR as determined by ECG | 1 minute

SECONDARY OUTCOMES:
Time of the first breath | 20 minutes
Time of regular breathing | 20 minutes
Mortality rate | 1 month (during hospitalization)
Number (%) of asphyxiated neonates | 5 min
Age at discharge/death (days) | 1 month

CONTACTS AND LOCATIONS:
Locations (2):
- St. Luke Catholic Hospital, Wolisso, Ethiopia, Addis Ababa, Ethiopia
- University of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cavallin F, Cori MS, Negash S, Azzimonti G, Vento G, Putoto G, Trevisanuto D. Heart Rate Determination in Newborns at Risk for Resuscitation in a Low-Resource Setting: A Randomized Controlled Trial. J Pediatr. 2020 Jun;221:88-92.e1. doi: 10.1016/j.jpeds.2020.02.026. Epub 2020 Mar 25. PMID 32222255